CLINICAL TRIAL: NCT01818115
Title: A Prospective, Multi-Center, Randomized Controlled Trial to Evaluate the Safety and Effectiveness of the Hydrus Implant for Lowering Intraocular Pressure in Glaucoma Patients Undergoing Cataract Surgery.
Brief Title: Safety and Efficacy Trial to Evaluate the Hydrus(TM) Implant in Subjects Undergoing Cataract Surgery.
Acronym: Hydrus II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ivantis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CP-10-001
Record Dates: First submitted 2012-02-29; First posted 2013-03-26 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Primary Open Angle Glaucoma; Glaucoma, Open Angle, Pseudo-exfoliative; Cataract Unilateral Pending Extraction
Keywords: POAG; PXG; IOL Surgery; CE Surgery
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- IOL placement with Hydrus Implant (Experimental): Cataract extraction with intraocular lens (IOL) placement and Hydrus Implant
  Interventions: Device: Hydrus Implant
- IOL placement only. (Active Comparator): Cataract Extraction with IOL placement only.
  Interventions: Procedure: IOL placement

INTERVENTIONS:
Device: Hydrus Implant
  Arms: IOL placement with Hydrus Implant
Procedure: IOL placement
  Arms: IOL placement only.

SUMMARY:
The objective of this study is to demonstrate the ability of the Hydrus Implant to lower intraocular pressure in glaucoma patients undergoing cataract surgery.

DETAILED DESCRIPTION:
This is a post-market, prospective, single-masked, randomized, controlled, multicenter clinical trial comparing Cataract Extraction (CE) surgery + Hydrus Implant vs CE surgery alone for the reduction of intraocular pressure (IOP) in patients with a positive diagnosis for open angle glaucoma (POAG) or pseudoexfoliative glaucoma. Eligible patients will be scheduled for cataract surgery. At the time of the procedure, qualified subjects will be randomized into 1 of 2 treatment groups: Hydrus Implant with cataract surgery or cataract surgery alone. Post-operative follow up will be conducted at regular intervals.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Primary Open Angle Glaucoma or Pseudoexfoliative Glaucoma.
* Operable, age-related cataract eligible for phacoemulsification.

Exclusion Criteria:

* Closed Angle and narrow angle forms of Glaucoma.
* Other Secondary Glaucoma, (such as neovascular, uveitic, traumatic, steroid induced, lens induced); glaucoma associated with increase episcleral venous pressure; congenital or developmental glaucoma.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-01; Primary Completion 2015-08 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Difference in proportion of subjects with 20% reduction in mean diurnal Intraocular Pressure (IOP) at 24 months following the wash-out of all glaucoma medications. | 24 months
  The 24 month diurnal IOP will be compared to the baseline value and a % change will be determined for each subject. A 20% drop in diurnal IOP is a successful response to treatment.

SECONDARY OUTCOMES:
Reduction in mean washed out IOP at 24 months | 24 months
  The mean diurnal IOP for each subject will be calculated and the sorted by group. The group average IOP will be compared to in-group baseline and between groups at the follow up time point.
Change in Best-corrected Visual Acuity (BCVA) from baseline to 12 months as measured by Early Treatment Diabetic Retinopathy Study (ETDRS) eye chart. | 12 months
  A 24 month visit will be conducted to confirm 12 month findings.
The proportion of eyes with IOP >5 mmHg to ≤19 mmHg following terminal washout. | 12 months
  A 24 month visit will be conducted to confirm 12 month findings.
Diurnal IOP at 12 months following washout | 12 months
  A 24 month visit will be conducted to confirm 12 month findings

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Norbert Pfeiffer, MD, Principal Investigator — Universitatsmedizin Mainz
Locations (7):
- Germany (2):
  - See Central Contact, Frankfurt
  - See Central Contact, Mainz
- Italy (2):
  - See Central Contact, Parma
  - See Central Contact, Torino
- See Central Contact, Rotterdam, Netherlands
- Spain (2):
  - See Central Contact, Madrid
  - See Central Contact, Zaragoza

IPD SHARING:
Plan to Share IPD: No